CLINICAL TRIAL: NCT02936778
Title: Risk Factors for Intensive Care Admission of Children With Severe Acute Wheeze or Asthma (SAA)
Brief Title: Status Asthmaticus on the Intensive Care Prospective - STATIC PRO
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Radboud University Medical Center (Other); Maasstad Hospital (Other); Amsterdam UMC, location VUmc (Other); UMC Utrecht (Other); University Medical Center Groningen (Other); Amphia Hospital (Other); Rijnstate Hospital (Other); Tergooi Hospital (Other); Maastricht University Medical Center (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Matthijs de Hoog, Prof. Dr., Erasmus Medical Center
Other Study IDs: NL52508.078.15
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Childhood Asthma With Status Asthmaticus
Keywords: Short-term medical and psychosocial functioning

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PICU (= case group): Children aged 2-18 years admitted to a Paediatric Intensive Care Unit in the Netherlands, with a diagnosis of acute wheeze or SAA.
- MC (= control group): Children aged 2-18 years admitted to a Medium Care in the Netherlands, with a diagnosis of acute wheeze or SAA.

SUMMARY:
This study will prospectively assess the impact and relevance of several risk factors for children with severe acute asthma (SAA) or acute wheeze that have been identified in retrospective studies. Secondary we will assess short-term medical and psychosocial functioning in patient (and parents) admitted to a PICU for SAA/acute wheeze versus a control group admitted to a MC for SAA/acute wheeze.

ELIGIBILITY:
Inclusion Criteria:

* Between 2 and 18 years of age
* Admission to a PICU for SAA or acute wheeze or admission to a MC for SAA or acute wheeze

Exclusion Criteria:

* Patient is outside of specified age range
* Down's Syndrome
* Congenital/acquired heart defect that interferes with normal SAA treatment
* Congenital/acquired airway defect (tracheomalacia/bronchomalacia)
* Primary/secondary immunodeficiency
* Pre-existing chronic pulmonary condition, known to mimic asthma: Cystic Fibrosis, Bronchopulmonary dysplasia, Bronchiolitis obliterans
* If both parents are not able to speak the Dutch language

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 2-18 years admitted to a Medium Care or Paediatric Intensive Care Unit in the Netherlands, with a diagnosis of acute wheeze or SAA.
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Undertreatment in children admitted to a PICU with a diagnosis of SAA/acute wheeze | Within the time of admission on the PICU/MC, preferably within 48 hours and during follow up after 3-6 months
  Undertreatment is defined as: Patient is not using inhaled corticosteroids (ICS), or Patient is using ICS < 7 days (counting from moment of admission to emergency department) according to treatment plan, or Patient is not using ICS according tot treatment plan.

SECONDARY OUTCOMES:
Exposure to triggers (single or combined) | Within the time of admission on the PICU/MC, preferably within 24 hours
  Pollution/airborne particulate matter (PM10), sensitization/allergen exposure, cigarette smoke exposure (measured by cotinine in urine), presence and type of virus in upper airway tract
Socio-economic status | Within the time of admission on the PICU/MC
Frequency of previous asthma-related hospital admissions and/or PICU admissions. | Within the time of admission on the PICU/MC and during follow up after 3-6 months
Severity of disease, defined using the GINA criteria for stepwise management of asthma. | Within the time of admission on the PICU/MC, preferably within 48 hours and during follow up after 3-6 months
Distribution of ADRB2-receptor polymorphisms compared to non-SAA population. | Through study completion, preferably within the time of admission on the PICU/MC

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands